CLINICAL TRIAL: NCT05473689
Title: Outcomes Post Treatment: Impact on Motor Impairment of Sleep Efficiency in SCI (OPTIMISE SCI Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-6214
Record Dates: First submitted 2022-07-19; First posted 2022-07-26 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries; Spine Disease
Keywords: sleep apnea; sleep-related breathing disorders
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Diseases; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Early-CPAP therapy group (Experimental): Individuals diagnosed with moderate-to-severe sleep-related breathing disorders (SRBDs) who will start CPAP therapy within the first 6 weeks after SCI.
  Interventions: Device: Continuous positive airway pressure (CPAP) therapy
- Delayed-CPAP therapy group (Active Comparator): Individuals diagnosed with moderate-to-severe SRBDs who will start on CPAP therapy at the 5th month after SCI.
  Interventions: Device: Continuous positive airway pressure (CPAP) therapy
- Non-CPAP therapy group (No Intervention): Individuals who are diagnosed with no or mild SRBD.

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) therapy — Continuous positive airway pressure (CPAP) therapy for moderate-to-severe sleep-related breathing disorders.
  Arms: Delayed-CPAP therapy group; Early-CPAP therapy group

SUMMARY:
This randomized clinical trial will compare three groups of individuals with cervical/thoracic, complete or incomplete spinal cord injury (SCI) that will undergo: (i) early CPAP therapy in the management of moderate-to-severe sleep-related breathing disorders (SRBDs) among adults at 6 weeks after SCI; (ii) delayed CPAP therapy in the management of moderate-to-severe SRBDs among adults at 22 weeks after SCI; and (iii) no treatment as they either have mild or no SRBD.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking adults (18 years of age or older)
* Acute (≤ 30 days after injury), cervical/thoracic (injury level at C2 to T12), complete or incomplete (AIS A to D) SCI
* Not being treated for sleep apnea prior to the spinal cord impairment onset.

Exclusion Criteria:

* Non-traumatic spinal cord disease at risk for neurologic progression (e.g., demyelinating spine diseases such as neuromyelitis optica and multiple sclerosis, spinal cord malignancy)
* Concomitant diseases of the central nervous system
* Preinjury chronic pain
* Other pre-existing diseases of the central nervous system
* Significant psychiatric disorders with recent episode of exacerbation
* Neuromuscular diseases
* Current substance misuse
* Known history of primary hypersomnia or secondary hypersomnia of any cause except for SRBDs (e.g., hypothyroidism, moderate or severe iron deficiency anemia, infections, depression, kidney failure, chronic fatigue syndrome, neurodegenerative diseases, and myotonic dystrophy)
* Epilepsy
* Vitamin B12 deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in International Standards for Neurological Classification of SCI (ISNCSCI) motor subscore from baseline to 6 months after recruitment | From baseline to 6 months after recruitment
  Motor assessment of muscles in the upper and lower extremities (100: normal; 0: complete paresis)
Change in International from baseline to 6 months after recruitment Standards for Neurological Classification of SCI (ISNCSCI) sensory subscore | From baseline to 6 months after recruitment
  Sensory assessment of dermatomes in the upper and lower extremities (224: normal; 0: no sensory function)
Change in Spinal Cord Independence Measure (SCIM) - version III - score from baseline to 6 months after recruitment | From baseline to 6 months after recruitment
  The SCIM scores varies from 0 to 100 and includes the following subscores: self-care (0-20); respiration and sphincter management (0-40); mobility (0-40).

SECONDARY OUTCOMES:
Change in Fatigue Severity Scale (FSS) from baseline to 6 months after recruitment | From baseline to 6 months after recruitment
  The FSS scores vary from 9 (normal) to 56 (the most severe degree of fatigue)
Change in Depression, Anxiety & Stress Scales- 21 (DASS-21) score from baseline to 6 months after recruitment | From baseline to 6 months after recruitment
  The DASS-21 scores vary from 0 (normal) to 42 (most severe symptoms of depression, anxiety and stress).
Change in Patient Health Questionnaire (PHQ-9) score from baseline to 6 months after recruitment | From baseline to 6 months after recruitment
  The PHQ-9 scores vary from 0 to 27, which means: 0-4 is the normal or minimal; 5-9 if the person is mildly depressed; 10-14 if the person is moderately depressed; 15-19 if the person has moderately severe depression; and 20-27 if the person is severely depressed.
Change in Medical Outcomes Study Sleep Scale (MOS-SS) from baseline to 6 months after recruitment | From baseline to 6 months after recruitment
  Scores for the sleep disturbance, snoring, respiratory problems, sleep adequacy, and daytime somnolence dimensions range from 0 (normal) to 100.
Change in Montreal Cognitive Assessment (MoCA test) score from baseline to 6 months after recruitment | From baseline to 6 months after recruitment
  The MoCA test scores vary from 0 to 30 (normal).

CONTACTS AND LOCATIONS:
Overall Officials: Julio C Furlan, MD, FRCPC, Principal Investigator — KITE Research Institute, University Health Network
Locations (1):
- KITE Toronto Research Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The UHN REB needs to approve any plan to share data from this RCT.

REFERENCES:
- [Derived] Furlan JC, Yao C, McKay M, Walsh S, Boulos M. Study protocol for the Outcomes Post-Treatment: Impact on Motor Impairment of Sleep Efficiency in Spinal Cord Injury (OPTIMISE SCI) - a randomised controlled trial. BMJ Open. 2025 Jun 6;15(6):e099266. doi: 10.1136/bmjopen-2025-099266. PMID 40480676